CLINICAL TRIAL: NCT03059745
Title: Evolution of Robotic Cholecystectomy; the U.C. Davis Experience.
Brief Title: Use of Robotics for Cholecystectomy; Retrospective Review of Outcomes, Set Up and Learning Curves
Status: Completed | Type: Observational
Sponsor: University of California, Davis (Other)
Responsible Party: Sponsor
Other Study IDs: 237231
Record Dates: First submitted 2014-01-27; First posted 2017-02-23 (Actual); Last update posted 2019-06-11 (Actual); Status verified 2019-06

CONDITIONS: Cholecystitis; Cholelithiasis
Keywords: Cholecystitis; Cholelithiasis
MeSH Terms: conditions — Cholecystitis; Cholelithiasis | interventions — Cholecystectomy

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Cholecystitis: Patients consented for robotic assisted cholecystectomy evaluated in study.
  Interventions: Procedure: Cholecystectomy

INTERVENTIONS:
Procedure: Cholecystectomy — Single Port and Multi-Port approaches trans-laparoscopic approaches with or without the use of the daVinci Surgical Robotic System.
  Other Names: daVinci Surgical Robotic System

SUMMARY:
Comparing the use of surgical robotics during a Cholecystectomy, comparing different platforms and approaches (multi port verses single port).

DETAILED DESCRIPTION:
This study is a restrospective review of charts, including operating room notes as well as operating room documentation of procedures. Currently there are numerous methods considered to be the Standard of Care in the surgical treatment of Cholecystitis, or Cholelithiasis, including Open Surgery, Laparoscopic, and Robotic Assisted Laparoscopic Surgery. This study retrospectively reviews the intraoperative and post operative clinical outcomes of Laparoscopic and Robotic Assisted Surgery at U.C. Davis Medical Center to: 1) establish the role of robotics in laparoscopic surgery, and 2) to assess the learning curve by surgeons.

ELIGIBILITY:
Inclusion Criteria:

* Patients that have undergone robotic assisted laparoscopic cholecystectomy

Exclusion Criteria:

* Patients under the age of 18, or not choosing to have surgery.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients which have undergone a robotic assisted laparoscopic cholecystectomy
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2004-06; Primary Completion 2017-03-03 (Actual); Study Completion 2017-03-03 (Actual)

PRIMARY OUTCOMES:
Comparing hernia rates between multi-port verses single port approaches. | June 2004 through May 2015
  Comparing multi port and single port approaches. Patients will be followed up under the standard of care model, normal clinical follow-ups required post surgery (10 Days to 2 weeks post operative) with additional clinical visits as required to monitor post operative complications (if any).

CONTACTS AND LOCATIONS:
Overall Officials: Tamas Vidovszky, MD, Principal Investigator — University of California, Davis
Locations (2):
- United States (2):
  - University of California Davis Health System, Sacramento, California
  - Univesity of California Davis Health System, Sacramento, California

IPD SHARING:
Plan to Share IPD: No